CLINICAL TRIAL: NCT02833831
Title: A Double-blind, Double-dummy, Randomized, 3-Period Cross-over, Placebo- and Positive Controlled Study to Evaluate the Effect of ALS-008176 on Cardiac Repolarization Interval in Healthy Subjects
Brief Title: Study to Evaluate the Effect of ALS-008176 on Cardiac Repolarization Interval in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR108169; 64041575RSV1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-06-21; First posted 2016-07-14 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — 4'-chloromethyl-2'-deoxy-3',5'-di-O-isobutyryl-2'-fluorocytidine; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (9):
- Part 1: Group 1 (Experimental): Participants will receive Treatment A (a single dose of ALS-008176 1,500 mg) or Treatment B (a single dose of placebo) under fasted conditions.
  Interventions: Drug: ALS-008176; Drug: Placebo
- Part 1: Group 2 (Experimental): Participants will receive Treatment C (a single dose of ALS-008176 2,500 mg) or Treatment D (a single dose of placebo) under fasted conditions.
  Interventions: Drug: ALS-008176; Drug: Placebo
- Part 1: Group 3 (Experimental): Participants will receive Treatment E (a single dose of ALS-008176 3,000 mg) or Treatment F (a single dose of placebo) under fasted conditions.
  Interventions: Drug: ALS-008176; Drug: Placebo
- Part 2: Sequence GHI (Experimental): Participants will receive Treatment G (a single dose of ALS-008176 3,000 mg + a single dose of moxifloxacin placebo under fasted conditions) then Treatment H (a single dose of ALS-008176 placebo + a single dose of moxifloxacin 400 mg under fasted conditions) then Treatment I (a single dose of ALS-008176 placebo + a single dose of moxifloxacin placebo under fasted conditions). There will be a washout period of at least 14 days between subsequent treatments.
  Interventions: Drug: ALS-008176; Drug: Placebo; Drug: Moxifloxacin
- Part 2: Sequence HIG (Experimental): Participants will receive Treatment H then Treatment I and then Treatment G. There will be a washout period of at least 14 days between subsequent treatments.
  Interventions: Drug: ALS-008176; Drug: Placebo; Drug: Moxifloxacin
- Part 2: Sequence IGH (Experimental): Participants will receive Treatment I then Treatment G and then Treatment H. There will be a washout period of at least 14 days between subsequent treatments.
  Interventions: Drug: ALS-008176; Drug: Placebo; Drug: Moxifloxacin
- Part 2: Sequence IHG (Experimental): Participants will receive Treatment I then Treatment H and then Treatment G. There will be a washout period of at least 14 days between subsequent treatments.
  Interventions: Drug: ALS-008176; Drug: Placebo; Drug: Moxifloxacin
- Part 2: Sequence HGI (Experimental): Participants will receive Treatment H then Treatment G and then Treatment I. There will be a washout period of at least 14 days between subsequent treatments.
  Interventions: Drug: ALS-008176; Drug: Placebo; Drug: Moxifloxacin
- Part 2: Sequence GIH (Experimental): Participants will receive Treatment G then Treatment I and then Treatment H. There will be a washout period of at least 14 days between subsequent treatments.
  Interventions: Drug: ALS-008176; Drug: Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: ALS-008176 — Participants will receive a single dose of ALS-008176 orally.
Drug: Placebo — Matching Placebo will be administered.
Drug: Moxifloxacin — Participants will receive a single dose of moxifloxacin 400 mg.
  Arms: Part 2: Sequence GHI; Part 2: Sequence GIH; Part 2: Sequence HGI; Part 2: Sequence HIG; Part 2: Sequence IGH; Part 2: Sequence IHG

SUMMARY:
The primary objective of this study is to evaluate the effect of supratherapeutic exposures of ALS-008176 on the QT/ corrected QT interval (QTc) interval in healthy participants (Panel 2).

DETAILED DESCRIPTION:
This is a two-part Phase 1 study consisting of a dose escalation part (Part 1) and a TQT part (Part 2), performed in two separate panels (Panels 1 and 2). Panel 1 will be a double blind (neither the researchers nor the participants know what treatment the participant is receiving), randomized (study medication assigned to participants by chance), placebo controlled dose escalation study in healthy participants to determine the safety, tolerability and pharmacokinetics of ALS-008176 after administration of single doses of 1500 milligrams (mg), 2500 mg and 3000 mg under fasted conditions. The final dose to be used in the Panel 2 will be determined based on the results of this dose escalation part. An interim analysis will be conducted on Panel 1 to select the dose for Panel 2. Panel 2 will be a double blind, double dummy, randomized, 3 period crossover (the same medications provided to all participants but in different sequence), placebo and positive controlled study to evaluate the effect of ALS-008176 on the QT/QTc interval in healthy participants. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Each participant must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and is willing to participate in the study
* Participant must be willing and able to adhere to the prohibitions and restrictions specified in protocol
* A female participant must be of non-childbearing potential, defined as either: a) Postmenopausal- A postmenopausal state is defined as no menses for at least 12 months without an alternative medical cause and a serum follicle stimulating hormone (FSH) level in the postmenopausal range (> 40 International units per liter [IU/L] or International units/milliliter [mIU/mL]); b) Permanently sterile- Permanent sterilization methods include hysterectomy, bilateral salpingectomy, bilateral tubal occlusion/ligation procedures (without reversal operation), and bilateral oophorectomy
* During the study and for a minimum of one spermatogenesis cycle (defined as approximately 90 days) after receiving the (last dose of) study drug, a male participant: a) who is sexually active with a woman of childbearing potential must agree to use a barrier method of contraception (example, condom with spermicidal foam/gel/film/cream/suppository); b) who is sexually active with a pregnant woman must use a condom; c) must agree not to donate sperm
* Female partners of male participants must either be surgically sterilized, postmenopausal (amenorrhea for a minimum of 1 year) or, if of childbearing potential, must agree to use at least one of the following contraceptive methods for 90 days following the last dose of study drug: a nonhormonal intrauterine device with spermicide; contraceptive sponge with spermicide, diaphragm with spermicide, cervical cap with spermicide, or oral, implantable, transdermal, or injectable hormonal contraceptives
* A female participant must have a negative serum beta human chorionic gonadotropin (b-hCG) pregnancy test at screening and on Day -1
* A female participant must agree not to donate eggs (ova, oocytes) during the study and for at least 90 days after receiving the (last dose of) study drug
* Participants must have a body mass index (BMI); weight (kilogram [kg])/height^2 (meter [m]^2) between 18.0 and 30.0 kg/m^2 (inclusive) at screening
* Participants must have a blood pressure (supine after at least 5 minutes rest) between 90 and 140 millimeters of Mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic at screening
* Participants must have a 12-lead electrocardiogram (ECG) consistent with normal cardiac conduction and function at screening, including: a) Sinus rhythm (heart rate between 45 and 100 beats per minute (bpm), inclusive); b) QT interval corrected for heart rate according to Fridericia (QTcF) interval between 350 milliseconds (ms) and 430 ms for male participants, and between 350 ms and 450 ms for female participants (inclusive); c) QRS interval of <110 ms; d) PR interval <=200 ms; e) Morphology consistent with healthy cardiac conduction and function
* Participants must be non-smokers for at least 3 months prior to screening
* Participants must be healthy on the basis of a medical evaluation that reveals the absence of any clinically significant abnormality and includes a complete physical examination, medical and surgical history, vital signs, ECGs, and the results of blood biochemistry and hematology tests and a urinalysis performed at screening. If there are abnormalities the participant may be included only if the Investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the Investigator
* Participants must have normal values for alanine aminotransferase (ALT) and aspartate aminotransferase (AST) (<= 1.0*upper limit of laboratory normal range [ULN])

Exclusion Criteria:

* Participants has a history of current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the Investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Participants with one or more laboratory abnormalities at screening as defined in the Protocol
* Participants with a history of clinically relevant heart rhythm disturbances including atrial, junctional, re-entry, and ventricular tachycardias, heart blocks and incomplete and complete right and left bundle branch blocks
* Participants with unusual T wave morphology (such as bifid T wave) likely to interfere with QTc measurements
* Participants with a past history of heart arrhythmias (extra systolic beats or tachycardia at rest) or with a history of risk factors for Torsade de Pointes syndrome (for example, hypokalemia or family history of short/long QT syndrome, or sudden unexplained death at a young age [less than or equal to 40 years], drowning or sudden infant death in a first degree relative [that is, sibling, offspring, or biological parent])
* Participants with electrolyte abnormalities (hypokalemia, hypocalcemia, hypomagnesemia) of grade 2 or above within 21 days prior to the (first) intake of the study drug
* Participants with any skin condition likely to interfere with ECG electrode placement or adhesion
* Participants with a breast implant or a history of thoracic surgery likely to cause abnormality of the electrical conduction through thoracic tissues
* Participants with any history of clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, or urticaria
* Participants with a history of clinically significant drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy diagnosed in previous studies with experimental drugs
* Participants with presence of any febrile illness or symptoms of upper or lower respiratory tract infection in the 14 days before the (first) administration of study drugs
* Participant has taken any disallowed therapies as noted in Concomitant Therapy before the planned (first) intake of study drug
* Participant has a history of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-5) criteria within 5 years before screening or positive test result(s) for alcohol and/or drugs of abuse (including barbiturates, opiates, cocaine, amphetamines, methadone, benzodiazepines, methamphetamine, tetrahydrocannabinol, phencyclidine, and tricyclic antidepressants) at screening
* Participant has known allergies, hypersensitivity, or intolerance to ALS-008176, moxifloxacin or its excipients
* Participant has known allergy to heparin or history of heparin-induced thrombocytopenia
* Participant has donated blood or blood products or had substantial loss of blood (more than 500 milliliter) within 3 months before the (first) administration of study drug or intention to donate blood or blood products during the study
* Participant has received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 90 days before the planned (first) intake of study drug
* Participant is a woman who is pregnant or breastfeeding
* Participant is a man who plans to father a child while enrolled in this study or within 90 days after the (last) intake of study drug, or who is unwilling to use acceptable methods of contraception as outlined in Protocol
* Participant has a history of hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibody positive, or other clinically active liver disease, or tests positive for HBsAg or anti HCV at screening
* Participant has a history of human immunodeficiency virus type 1 (HIV-1) or HIV-2 infection, or tests positive for HIV-1 or -2 at screening
* The participant has preplanned surgery or procedures that would interfere with the conduct of the study
* Vulnerable participant (example, incarcerated individuals)
* Participant with lack of good/reasonable venous access
* Participant is an employee of the Investigator or study site with direct involvement in the proposed study or other studies under the direction of that Investigator or study site, or a family member of the employees or the Investigator, or an employee of the Sponsor
* Participant has any condition for which, in the opinion of the Investigator, participation would not be in the best interest of the participant (example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Participant has previously been dosed with ALS-008176 in more than 3 single-dose studies with ALS-008176
* Participant has previously been dosed with ALS-008176 in a multiple-dose study with ALS 008176

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2017-02-17 (Actual); Study Completion 2017-02-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Corrected QT intervals (QTc) | Baseline up to Day 2
  Change from baseline in QTc intervals with Fredericia correction will be analyzed.

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | 10 to 14 days after last study drug intake
Change from baseline in ECG parameters: RR interval, PR interval and QRS interval | Baseline up to Day 2
  Change from baseline in other ECG parameters (RR interval, PR interval and QRS interval) will be analyzed.
ALS-008112 and ALS 008144 plasma concentration-effect relationship for changes in QT/QTc (Panels 1 and 2) | up to Day 15 in Panel 1; up to Day 2 in Panel 2
Change from Baseline in QT/QTc interval in healthy subjects (Panel 2) | up to Day 2
Maximum Observed Plasma Concentration (Cmax) | up to Day 15 in Panel 1; up to Day 2 in Panel 2
Time to Reach Maximum Observed Plasma Concentration (Tmax) | up to Day 15 in Panel 1; up to Day 2 in Panel 2
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0- last]) | up to Day 15 in Panel 1
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0- infinity]) | up to Day 15 in Panel 1
Elimination Half-Life (t1/2) | up to Day 15 in Panel 1
Elimination Rate Constant (Lambda[z]) | up to Day 15 in Panel 1
Plasma Concentration at 24 hours post dosing | up to Day 15 in Panel 1
Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours (AUC[0-24]) | up to Day 15 in Panel 1; up to Day 2 in Panel 2
Change from baseline in Heart Rate | Baseline up to Day 2
  Change from baseline in heart rate will be analyzed.
Change from baseline in T wave morphology | Baseline up to Day 2
  Change from baseline in T wave morphology will be analyzed.
Frequency of T wave morphology changes | up to Day 2
  T-wave morphology changes will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Tempe, Arizona, United States